CLINICAL TRIAL: NCT02962791
Title: Prospective Randomized Trial Comparing TRIPLE Site ventriculAr Stimulation Versus Conventional Pacing in CRT canDidates: TRIPLEAD Trial
Brief Title: Prospective Randomized Trial Comparing TRIPLE Site ventriculAr Stimulation Versus Conventional Pacing in CRT canDidates
Acronym: TRIPLEAD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Rouen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2016/091/HP
Record Dates: First submitted 2016-11-09; First posted 2016-11-11 (Estimated); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Cardiac Resynchronization Therapy
Keywords: symptomatic heart failure
MeSH Terms: interventions — Echocardiography

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Stimulation of 3 ventricular sites (Experimental): Cardiac resynchronization therapy implantation wil be done as usual, except the additional stimulation lead. Standard Echocardiography will be done at one year
  Interventions: Procedure: Cardiac resynchronization therapy implantation; Device: Stimulation of 3 ventricular sites; Device: Echocardiography
- Stimulation of 2 ventricular sites (Active Comparator): Cardiac resynchronization therapy implantation wil be done as usual. Standard Echocardiography will be done at one year
  Interventions: Procedure: Cardiac resynchronization therapy implantation; Device: Stimulation of 2 ventricular sites; Device: Echocardiography

INTERVENTIONS:
Procedure: Cardiac resynchronization therapy implantation — Cardiac resynchronization therapy implantation will be done for patient with symptomatic heart failure
Device: Stimulation of 3 ventricular sites — Cardiac resynchronization therapy with stimulation of 3 ventricular sites
  Arms: Stimulation of 3 ventricular sites
Device: Stimulation of 2 ventricular sites — Cardiac resynchronization therapy with stimulation of 2 ventricular sites
  Arms: Stimulation of 2 ventricular sites
Device: Echocardiography — Standard Echocardiography will de bone for patient

SUMMARY:
Cardiac resynchronization therapy (CRT) is a recommended treatment for selected patients with symptomatic heart failure (HF). Although most treated patients show a benefit from CRT, a lack of response is observed for about 25-30% of them whatever the response criteria used either based on the clinical status (NYHA class, Packer clinical composite score) or on ventricular remodeling parameters assessed by echography (Left ventricle end of systole volume). This rate has remained remarkably stable since the therapy started and has motivated many studies to better understand the underlying physiopathology and the CRT action mechanisms.

Among the various research axes to improve CRT response and responders rate, increasing the number of pacing sites in an attempt to better homogenize the cardiac mechanical activity has been evaluated. A configuration with two RV leads and one LV lead was tested acutely in three studies. In all cases, it demonstrated a significant improvement of cardiac performance whether assessed by echographic parameters or LV dp/dt measurements. Additionally feasibility of this approach for long term CRT delivery was demonstrated during a previous study. First results with triple-site ventricular stimulation are encouraging and its clinical efficacy should now be tested on a larger population in order to conclude on its interest for CRT candidates.

ELIGIBILITY:
Inclusion Criteria:

* Patient who signed the MEC approved informed consent
* Patient older than 18
* Patient with a CRT (CRT-P or D) indication as per ESC guidelines 2013
* Left Ventricular Ejection Fraction (LVEF) ≤ 35%
* NYHA class II/III/IV despite optimal medical treatment
* Left Bundle Branch Block (LBBB) and QRS ≥ 120 ms (class IA and IB indications) or in the absence of LBBB QRS > 150 ms (class IIA indication)
* De novo implantation
* Sinus rhythm

Exclusion Criteria:

* Permanent supra ventricular tachycardia
* Pacing indication for 3rd degree AV block
* Impossibility to perform FU at the investigative center
* Pregnancy
* Adults under legal protection
* Heart transplant candidates
* Concomitant pathology that may interfere with the study results

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2017-10-24 (Actual); Primary Completion 2020-11-20 (Actual); Study Completion 2020-11-20 (Actual)

PRIMARY OUTCOMES:
Difference from baseline in Left Ventricular End-Systolic Volume | 12 months
  Left Ventricular End-Systolic Volume will be evaluated using echocardiography

SECONDARY OUTCOMES:
Difference from baseline in left ventricular remodelling | 12 months
  Left ventricular remodelling will be evaluated using echocardiography
Number of patients alive | 12 months
Number of adverse events | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Frédéric ANSELME, Pr, Principal Investigator — University Hospital, Rouen
Locations (1):
- Rouen University Hospital, Rouen, France

IPD SHARING:
Plan to Share IPD: No